CLINICAL TRIAL: NCT06274736
Title: Post-marketing Cohort Study to Confirm the Safety and Performance of Motiva® Sizers in Breast Augmentation and Reconstruction Procedures
Brief Title: Safety and Performance of Motiva® Sizers
Status: Recruiting | Type: Observational
Sponsor: Establishment Labs (Industry)
Responsible Party: Sponsor
Other Study IDs: CLINP-001012
Record Dates: First submitted 2023-12-27; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Breast Implant; Complications; Breast Implantation; Methods, Safety and Performance; Mammaplasty; Breast Reconstruction; Breast Augmentation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Women who will undergo a breast augmentation or reconstruction with Motiva® Sizer during surgery.
  Interventions: Device: Motiva Sizer
- Women who will undergo a breast augmentation or reconstruction without Motiva® Sizer during surgery.

INTERVENTIONS:
Device: Motiva Sizer — No intervention will be made,
  Groups: Women who will undergo a breast augmentation or reconstruction with Motiva® Sizer during surgery.

SUMMARY:
The Motiva® Sizer clinical study is a four-year, multicenter, post-marketing, and cohort study, designed to confirm the safety and performance of Motiva® Sizer in breast augmentation or reconstruction procedures.

The research will include 330 women, divided into two groups of 165 participants each (150 breast augmentation participants and 15 reconstruction participants). The Motiva® Sizer exposed group will consist of women who will undergo breast augmentation or reconstruction surgery with the use of Motiva® Sizer during the procedure, and a non-exposed group will consist of women who will undergo breast augmentation or reconstruction surgery without the use of Motiva® Sizer. This study will be conducted in Costa Rica.

The main goal is to evaluate the safety and the performance of the Motiva® Sizer. To this end, the results of both groups will be compared in terms of surgical complications, surgeon's, and participant's satisfaction level as well as reoperation rates.

After the augmentation or reconstruction surgery, participants will be scheduled for the following follow-up visits, (1) between 3 and 7 postoperative days, (2) between 3 and 6 postoperative weeks, (3) at 3 and (4) 6 postoperative months, and (5, 6 and 7) annually thereafter for a period of three consecutive years. In case any participant has an adverse event due to the procedure, and if required by the physician, an additional visit will be made to assess her, and this information as well as that of the scheduled visits should be recorded in the electronic data collection notebook.

ELIGIBILITY:
Inclusion Criteria:

* Female, 18 years of age or older.
* The participant will be undergoing a breast augmentation or reconstruction procedure.
* To possess enough and adequate tissue to cover the implants.
* Willingness to comply with all study requirements, including signing the informed consent document and agreeing to attend all required follow-up visits.

Exclusion Criteria:

* Existing rib injuries.
* Inadequate or unsuitable tissue for augmentation or reconstruction surgery at the physician's discretion.
* History of abscesses or infections in the breast area.
* Current pregnancy or breastfeeding, or full-term pregnancy or breastfeeding in the six months prior to enrollment.
* History of sensitivity to silicone.
* Any medical condition, such as underweight or obesity, diabetes, autoimmune disease or severe chronic pulmonary or cardiovascular disease, psychological/psychiatric disorders that may result in unduly high surgical risk and/or significant postoperative complications.
* Active or recurrent breast cancer.
* Consumption of any medication that, in the investigator's experience, may pose an increased risk of complications or interfere with wound healing ability, such as corticosteroid therapy or blood clotting medication (e.g., concomitant treatment with warfarin).
* Not living in the country where the procedure was performed , which prevents him/her from attending follow-up visits .

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women over 18 years of age who will undergo breast augmentation or reconstruction. They will be divided into two groups:
  * Group exposed to Motiva® Sizer: 165 participants (150 breast augmentation participants and 15 reconstruction participants).
  * Group not exposed to Motiva® Sizer: 165 participants (150 breast augmentation participants and 15 reconstruction participants).
Sampling Method: Non-Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2023-04-10 (Actual); Primary Completion 2027-04-10 (Estimated); Study Completion 2027-07-10 (Estimated)

PRIMARY OUTCOMES:
Motiva Sizers Safety (complications) | 3 years
  Cumulative incidence of complications between participants in whom Motiva® Sizer was used during breast augmentation or reconstruction surgery, and participants in whom intraoperative breast sizers were not used during breast augmentation or reconstruction surgery
Motiva Sizers Performance (satisfaction) | 3 years
  Percentage of participants and surgeons who are satisfied or very satisfied with surgery´s results with and without Motiva® Sizer. (based on 5-point Likert scale, in which 1 is Very dissatisfied, 2 Dissatisfied, 3 Neither satisfied nor dissatisfied, 4 Satisfied, 5 Very satisfied) measured at 3rd, 6th months after surgery and 1st, 2nd and 3rd year.

SECONDARY OUTCOMES:
Motiva Sizers Safety (reoperations) | 3 years
  Re-operation rates between participants in whom Motiva® Sizers were used during augmentation or breast reconstruction surgery and participants in whom Motiva® Sizers were not used during augmentation or breast reconstruction surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Establishment Labs, Coyol, Alajuela Province, Costa Rica